CLINICAL TRIAL: NCT02691845
Title: Initiating and Maintaining Physical Activity in Depressed Individuals
Acronym: Project MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL127695 (NIH); R56HL127695 (NIH); R01HL127695 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-02-25 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Crisis Intervention; Helium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BA (Other): Brief advice to exercise. This serves as a control condition.
  Interventions: Behavioral: BA (brief advice)
- BA + SHE + HE (Active Comparator): Brief advice to exercise + supervised & home-based exercise + health education
  Interventions: Behavioral: BA (brief advice); Behavioral: SHE (supervised and home-based exercise); Behavioral: HE (health education)
- BA + SHE + CBEX (Experimental): Brief advice to exercise + supervised & home-based exercise + cognitive-behavioral sessions focused on increasing and maintaining exercise
  Interventions: Behavioral: BA (brief advice); Behavioral: SHE (supervised and home-based exercise); Behavioral: CBEX (cognitive-behavioral sessions focused on increasing and maintaining exercise)

INTERVENTIONS:
Behavioral: BA (brief advice)
Behavioral: SHE (supervised and home-based exercise)
  Arms: BA + SHE + CBEX; BA + SHE + HE
Behavioral: HE (health education)
  Arms: BA + SHE + HE
Behavioral: CBEX (cognitive-behavioral sessions focused on increasing and maintaining exercise)
  Arms: BA + SHE + CBEX

SUMMARY:
The investigators propose a randomized clinical trial in which 240 depressed individuals are assigned to one of three arms, with each successive arm having an added component that may serve to increase and maintain physical activity:

1. brief advice (BA) to exercise (control condition);
2. BA + supervised & home-based exercise (SHE) + health education (HE) contact control; and
3. BA + SHE+ cognitive-behavioral sessions focused on increasing and maintaining exercise (CBEX).

The primary aim is to assess and optimize the safety, feasibility, acceptability of each intervention component, as well as barriers limiting their effectiveness in order to prepare for a larger scale randomized clinical trial.

DETAILED DESCRIPTION:
The investigators propose a randomized clinical trial in which 240 depressed individuals are assigned to one of three arms, with each successive arm having an added component that may serve to increase and maintain physical activity:

1. brief advice (BA) to exercise (control condition);
2. BA + supervised & home-based exercise (SHE)+health education (HE) contact control; and
3. BA+SHE+ cognitive-behavioral sessions focused on increasing and maintaining exercise (CBEX).

There are two phases for participants: intervention phase (3 months), which consists of intensive contact, and the follow-up phase (6 months). BA will consist of one, 45-minute session about public health recommendations, and strategies for getting started. SHE will be a 12-week intervention consisting of 1x/week supervised exercise plus exercise prescriptions for home-based exercise with the goal of gradually achieving the public health recommendation of 150 minutes/week of moderate-to-vigorous physical activity (MVPA), CBEX and HE sessions will be individual, 30-minute, weekly sessions during the intervention phase. CBEX will address barriers to physical activity that are particularly pronounced in depression -i.e., anhedonia, decreased motivation, and decreased energy, as well as poor problem-solving skills. During the follow-up phase, groups who received SHE during the intervention phase will receive brief, monthly phone check-ins from an exercise specialist.

Primary Aims:

1. To compare the efficacy of the 3 arms for increasing physical activity during the 12-week intervention phase. We hypothesize that BA + SHE + CBEX will be superior to BA + SHE + HE, and that BA + SHE + HE will be superior to BA alone in terms of objectively measured MVPA levels.
2. To compare the longer-term impact of the three arms on objectively-measured minutes of MVPA at 6- and 9-month follow-ups (i.e., follow-up phase). Hypotheses are the same as for the intervention phase (aim #1).

   Secondary Aims:
3. To assess the impact of proposed intervention combinations on depression, physical health outcomes including cardiorespiratory fitness and body composition, and self-reported MVPA in all phases. Hypotheses mirror those described in our primary aims above.
4. To determine whether amount of MVPA mediates the association between group assignment and change in depressive symptoms. We hypothesize that amount of MVPA will serve as a mediator.
5. To examine behavior change theory-based mediators of the association between group assignment and MVPA. Hypothesized mediators include: perceived benefits of exercise, perceived barriers to exercise, exercise self-efficacy, intrinsic motivation to exercise, and identified motivation to exercise.
6. To examine whether social and environmental barriers to exercise predict exercise maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary, i.e., have not participated regularly in moderate-to-vigorous physical activity (MVPA) for 90 minutes per week or more for more than 6 weeks of the past 12 weeks.
2. Medically cleared for MVPA, documented by a note from their primary care provider.
3. No significant medical condition or physical disability that would interfere with physical activity or study participation. The investigators will exclude individuals with significant cardiovascular disease, hematologic disorders, and autoimmune disorders. The investigators will also exclude individuals who are planning a surgery in the next 9 months and those with dementia.
4. Elevated depression symptoms. To meet criteria for elevated symptoms, participants must have a QIDS score of 8 or greater (i.e., at least moderate depression levels), and must have a score of "1" or greater on at least one of the two core DSM-V depressive symptoms, i.e., sad mood or anhedonia. -
5. No current bulimia or anorexia (past 3 months); no MDD with psychotic symptoms (past 6 months); no history of bipolar disorder, schizophrenia, or a chronic psychotic condition; (assessed using the SCID).
6. No hazardous drug or alcohol use in the past 6 months, as assessed by: a. no substance abuse treatment in the past 6 months; and b. does not meet criteria for a moderate or severe substance use disorder in the past 6 months.
7. Depression is not very severe, i.e., QIDS score is <= 20.
8. No suicidality requiring immediate treatment.
9. Not pregnant or planning on becoming pregnant in the next year.
10. Understands English sufficiently well to consent and complete study assessments.
11. Aged 18-65.
12. Able to make one of the 2 available exercise class times.
13. Able to walk 1 mile
14. Weight does not exceed 375 lbs.
15. If participants are aged 60 or older, or if there is any concern about their cognitive capacity, participants will undergo a brief cognitive functioning screener, the Montreal Cognitive Assessment (MOCA). Participants are required to achieve a score within 1 SD of the mean for their age and education level to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change in minutes of moderate-vigorous physical activity (MVPA) per week assessed via accelerometer | from baseline to 3 months, 6 months, 9 months

SECONDARY OUTCOMES:
change in depression assessed via Quick Inventory of Depression Symptoms | Baseline to 3 months, 6 months, 9 months
  depression assessed via blind evaluator using the Quick Inventory of Depression Symptoms (QIDS)
change in cardiorespiratory fitness | Baseline to 3 months, 6 months, 9 months
change in self-report of MVPA assessed via International physical activity questionnaire | Baseline to 3 months, 6 months, 9 months
change in Self-report of pain assessed via the SF-36 | Baseline to 3 months, 6 months, 9 months
change in Self-report of overall health assessed via the SF-36 | Baseline to 3 months, 6 months,9 months
change in Self-report of physical functioning assessed via the SF-36 | Baseline to 3 months, 6 months, 9 months
number, severity, impairment of adverse events | 3 months, 6 months, 9 months
change in anxiety assessed via state-trait anxiety inventory | Baseline to 3 months, 6 months, 9 months
change in irritability assessed via Brief irritability test | Baseline to 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital; Ana Abrantes, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No